CLINICAL TRIAL: NCT03901339
Title: Phase 3 Study of Sacituzumab Govitecan (IMMU-132) Versus Treatment of Physician's Choice (TPC) in Subjects With Hormonal Receptor-Positive (HR+) Human Epidermal Growth Factor Receptor 2 (HER2) Negative Metastatic Breast Cancer (MBC) Who Have Failed at Least Two Prior Chemotherapy Regimens
Brief Title: Study of Sacituzumab Govitecan-hziy Versus Treatment of Physician's Choice in Participants With HR+/HER2- Metastatic Breast Cancer
Acronym: TROPiCS-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-09; 2018-004201-33 (EudraCT Number)
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan-hziy (Experimental): Participants will receive sacituzumab govitecan-hziy 10 mg/kg via intravenous (IV) injection administered on Day 1 and Day 8 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Treatment of Physician's Choice (TPC) (Active Comparator): Participants will receive TPC determined prior to randomization from one of the following single-agent treatment:
  Dosing per National Comprehensive Cancer Network (NCCN) guidelines (with dose modifications for if toxic)
  * Eribulin: 1.4 mg/m^2 for North American sites, 1.23 mg/m^2 for European sites) via IV on Days 1 and 8 of a 21-day cycle
  * Capecitabine: 1000-1250 mg/m^2 orally twice daily for 2 weeks followed by a 1-week rest period given as a 21-day cycle
  * Gemcitabine: 800-1200 mg/m^2 via IV on Days 1, 8, and 15 of each 28-day cycle or per institution
  * Vinorelbine: 25 mg/m^2 via IV on Day 1 weekly cycle per institution
  Interventions: Drug: Eribulin; Drug: Capecitabine; Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; GS-0132
  Arms: Sacituzumab Govitecan-hziy
Drug: Eribulin — Administered intravenously per NCCN guidelines
  Arms: Treatment of Physician's Choice (TPC)
Drug: Capecitabine — Administered orally per NCCN guidelines
  Arms: Treatment of Physician's Choice (TPC)
Drug: Gemcitabine — Administered intravenously per NCCN guidelines
  Arms: Treatment of Physician's Choice (TPC)
Drug: Vinorelbine — Administered intravenously per NCCN guidelines
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
The primary objective of this study is to assess and compare the efficacy and safety of sacituzumab govitecan-hzi versus treatment of physician's choice (TPC) in participants with hormonal receptor-positive (HR+) human epidermal growth factor receptor 2 (HER2-) negative metastatic breast cancer (MBC).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented evidence of hormone receptor-positive human epidermal growth factor receptor 2 negative (HER2-negative) (hormonal receptor-positive (HR+)/HER2-) metastatic breast cancer (MBC) confirmed.
* Refractory to or relapsed after at least 2, and no more than 4, prior systemic chemotherapy regimens for metastatic disease:

  * At least 1 taxane in any setting.
  * At least 1 prior anticancer hormonal treatment in any setting.
  * At least 1 cyclin-dependent kinase inhibitor 4/6 in any setting.
* Eligible for one of the chemotherapy options listed in the TPC arm.
* Documented disease progression after the most recent therapy.
* Adequate bone marrow function (hemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1,500 per mm^3, platelets ≥ 100,000 per mm^3).
* Adequate renal function: calculated creatinine clearance ≥ 30 mL/minute according to the Cockcroft and Gault formula .
* Adequate liver function (bilirubin ≤ 1.5 institutional upper limit of normal (IULN), or ≤ 3 IULN for individuals with documented Gilbert's syndrome, aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x IULN (in the case of liver metastases ≤ 5.0 x IULN)).
* Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta human chorionic gonadotropin (ß-hCG)).

Key Exclusion Criteria:

* Previous treatment with topoisomerase 1 Inhibitors as a free form or as other formulations.
* History of significant cardiovascular disease or clinically significant electrocardiogram (ECG) abnormality.
* Active serious infection requiring antibiotics.
* Any medical or other condition which, in the opinion of the Investigator, causes the individual to be medically unfit to receive sacituzumab govitecan or unsuitable for any reason.
* Locally advanced MBC (stage IIIc) in individuals who are candidates for curative intent therapy at the time of study enrollment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (113):
- United States (55):
  - HonorHealth Research Institute, Avondale, Arizona
  - Arizona Oncology Associates, PC, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - University of California, Irvine Medical Center-Chao Family Comprehensive Cancer Center, Orange, California
  - Southern California Permanente Medical Group, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Yale University Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Inc., Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Mercy Medical Center, Medical Oncology & Hematology, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Allina Health, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Summit Medical Group, Florham Park, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Laura and Isaac Perlmutter Cancer Center/NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - The West Clinic, PC dba West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Houston Methodist Hospital/Houston Methodist Cancer Center, Houston, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - UT Health San Antonio - Mays Cancer Center, San Antonio, Texas
  - Virginia Cancer Specialists, Arlington, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. DBA Blue Ridge Cancer Care, Salem, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Belgium (4):
  - Chirec Cancer Institute, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Canada (3):
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Centre Hospitalier de L'Universite de Montreal - Hôpital Notre-Dame, Montreal
  - Centre Hospitalier Universitaire de Sherbrooke - Fleurimont, Sherbrooke
- France (10):
  - Hopital de Mercy, Ars-Laquenexy
  - Institut Sainte Catherine, Avignon
  - Hôpital Jean-Minjoz, Besançon
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
- Germany (14):
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Gynakologisches Zentrum Bonn, Bonn
  - Marienhospital Bottrop, Bottrop
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Essen
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt
  - Onkologische Schwerpunktpraxis Eppendorf, Hamburg
  - Gynakologisch-Onkologische Praxis Hannover, Hanover
  - DIAKOVERE Krankenhaus gGmbH Henriettenstift - Standort Kirchrode, Hanover
  - Nationales Centrum für Tumorerkrankungen - Heidelberg, Heidelberg
  - Praxisklinik für Hämatologie und Onkologie Koblenz, Koblenz
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum Mutterhaus der Borromäerinnen, Trier
- Italy (7):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale di Desio, Desio
  - Ospedale Vito Fazzi di Lecce, Lecce
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera San Gerardo di Monza, Monza
  - Azienda Unità Sanitaria Locale di Piacenza-Ospedale Guglielmo da Saliceto, Piacenza
  - IFO Istituto Nazionale dei Tumori Regina Elena, Rome
- Netherlands (3):
  - Antoni van Leeuwenhoekziekenhuis, Amsterdam
  - Medisch Centrum Haaglanden Antoniushove, Leidschendam
  - Maastricht UMC+, Maastricht
- Spain (11):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Quirónsalud Barcelona Instituto Oncologico Baselga, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Provincial de Castellón, Castillón
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Instituto Oncologico Bureau (IOB), Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (6):
  - Royal Cornwall Hospital NHS Trust, Cornwell
  - Royal Surrey County Hospital, Guildford
  - Leicester Royal Infirmary, Leicester
  - Barts Health NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Loirat D, Tredan O, Ciruelos E, Dalenc F, Gomez Pardo P, Jhaveri KL, Delaney R, Valdez T, Wang H, Motwani M, Yoon OK, Verret W, Tolaney SM. Overall survival with sacituzumab govitecan in hormone receptor-positive and human epidermal growth factor receptor 2-negative metastatic breast cancer (TROPiCS-02): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Oct 21;402(10411):1423-1433. doi: 10.1016/S0140-6736(23)01245-X. Epub 2023 Aug 23. PMID 37633306
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Loirat D, Tredan O, Ciruelos E, Dalenc F, Pardo PG, Jhaveri KL, Delaney R, Fu O, Lin L, Verret W, Tolaney SM. Sacituzumab Govitecan in Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Metastatic Breast Cancer. J Clin Oncol. 2022 Oct 10;40(29):3365-3376. doi: 10.1200/JCO.22.01002. Epub 2022 Aug 26. PMID 36027558
- [Background] Rugo HS, Bardia A, Tolaney SM, Arteaga C, Cortes J, Sohn J, Marme F, Hong Q, Delaney RJ, Hafeez A, Andre F, Schmid P. TROPiCS-02: A Phase III study investigating sacituzumab govitecan in the treatment of HR+/HER2- metastatic breast cancer. Future Oncol. 2020 Apr;16(12):705-715. doi: 10.2217/fon-2020-0163. Epub 2020 Mar 30. PMID 32223649
- [Background] Rugo HS, Schmid P, Tolaney SM, Dalenc F, Marme F, Shi L, Verret W, Shah A, Gharaibeh M, Bardia A, Cortes J. Health-related quality of life with sacituzumab govitecan in HR+/HER2- metastatic breast cancer in the phase III TROPiCS-02 trial. Oncologist. 2024 Sep 6;29(9):768-779. doi: 10.1093/oncolo/oyae088. PMID 38748596
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Spears PA, Tolaney SM. A plain language summary of the TROPiCS-02 study in patients with breast cancer (HR-positive/HER2-negative). Future Oncol. 2024 Apr;20(11):635-651. doi: 10.2217/fon-2023-0845. Epub 2024 Jan 25. PMID 38270051
- [Background] Rugo HS, Bardia A, Tolaney S. Sacituzumab govitecan for metastatic breast cancer: the TROPiCS-02 trial - Authors' reply. Lancet. 2024 Jul 27;404(10450):339-340. doi: 10.1016/S0140-6736(24)01049-3. No abstract available. PMID 39067902
- [Derived] McCann KE, Hurvitz SA. Innovations in targeted therapies for triple negative breast cancer. Curr Opin Obstet Gynecol. 2021 Feb 1;33(1):34-47. doi: 10.1097/GCO.0000000000000671. PMID 33093337
- [Derived] Kalinsky K, Diamond JR, Vahdat LT, Tolaney SM, Juric D, O'Shaughnessy J, Moroose RL, Mayer IA, Abramson VG, Goldenberg DM, Sharkey RM, Maliakal P, Hong Q, Goswami T, Wegener WA, Bardia A. Sacituzumab govitecan in previously treated hormone receptor-positive/HER2-negative metastatic breast cancer: final results from a phase I/II, single-arm, basket trial. Ann Oncol. 2020 Dec;31(12):1709-1718. doi: 10.1016/j.annonc.2020.09.004. Epub 2020 Sep 15. PMID 32946924
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=IMMU-132-09

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Belgium, Canada, France, Germany, Italy, the Netherlands, Spain, the United Kingdom, and the United States.
Pre-assignment Details: 776 participants were screened.
Groups:
- Sacituzumab Govitecan: Participants received sacituzumab govitecan 10 mg/kg of body weight, administered as a slow intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, occurrence of unacceptable adverse events (AEs), or another treatment discontinuation criterion was met (up to 40.1 months).
- Treatment of Physician's Choice (TPC): Participants received TPC (ie, eribulin, capecitabine, gemcitabine, or vinorelbine), administered as a single-agent treatment that was determined by the investigator before participant randomization until progression of disease, occurrence of unacceptable adverse events (AEs), or another treatment discontinuation criterion was met. Dosing per National Comprehensive Cancer Network (NCCN) guidelines (with dose modifications for if toxic)
  * Eribulin was administered IV at a dose 1.4 mg/m^2 at North American sites and 1.2 mg/m^2 at European sites on Days 1 and 8 of a 21-day cycle (up to 22.5 months).
  * Capecitabine 1000 to 1250 mg/m^2 was administered in a 21-day cycle, with capecitabine administered orally twice daily for 2 weeks followed by 1-week rest period (up to 12.9 months).
  * Gemcitabine 800 to 1200 mg/m^2 was administered IV on Days 1, 8, and 15 of a 28-day cycle (up to 22.3 months).
  * Vinorelbine 25 mg/m^2 was administered as a weekly IV injection (up to 8.1 months). Vinorelbine was not allowed as TPC for any participant with Grade 2 neuropathy.
Period: Overall Study
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Started | 272 | 271
Received at Least 1 Dose of Study Drug | 268 | 249
Completed | 0 | 0
Not Completed | 272 | 271
Not completed — Death | 220 | 192
Not completed — Informed consent withdrawn | 13 | 40
Not completed — Sponsor request | 30 | 23
Not completed — Reason not specified | 5 | 7
Not completed — Lost to Follow-up | 4 | 7
Not completed — Covid19 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population included all participants who were randomized, regardless of whether they received study treatment or not.
Groups:
- Sacituzumab Govitecan: Participants received sacituzumab govitecan 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, occurrence of unacceptable AEs, or another treatment discontinuation criterion was met (up to 40.1 months).
- Treatment of Physician's Choice (TPC): Participants received TPC (ie, eribulin, capecitabine, gemcitabine, or vinorelbine), administered as a single-agent treatment that was determined by the investigator before participant randomization until progression of disease, occurrence of unacceptable AEs, or another treatment discontinuation criterion was met. Dosing per NCCN guidelines (with dose modifications for if toxic)
  * Eribulin was administered IV at a dose 1.4 mg/m^2 at North American sites and 1.2 mg/m^2 at European sites on Days 1 and 8 of a 21-day cycle (up to 22.5 months).
  * Capecitabine 1000 to 1250 mg/m^2 was administered in a 21-day cycle, with capecitabine administered orally twice daily for 2 weeks followed by 1-week rest period (up to 12.9 months).
  * Gemcitabine 800 to 1200 mg/m^2 was administered IV on Days 1, 8, and 15 of a 28-day cycle (up to 22.3 months).
  * Vinorelbine 25 mg/m^2 was administered as a weekly IV injection (up to 8.1 months). Vinorelbine was not allowed as TPC for any participant with Grade 2 neuropathy.
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC) | Total~(N=543)
Number analyzed (Participants) | 272 | 271 | 543
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 199 | 204 | 403
  >=65 years | 73 | 67 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.5) | 56 (10.4) | 56 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 270 | 268 | 538
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 222 | 204 | 426
  Unknown or Not Reported | 44 | 55 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 184 | 178 | 362
  Race: Unknown or Not Reported | 69 | 70 | 139
  Race: Black or African American | 8 | 13 | 21
  Race: Asian | 11 | 5 | 16
  Race: Other or More Than One Race | 0 | 4 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 115 | 113 | 228
  France | 64 | 73 | 137
  Spain | 35 | 34 | 69
  Germany | 20 | 26 | 46
  Belgium | 16 | 9 | 25
  Italy | 9 | 6 | 15
  United Kingdom | 7 | 7 | 14
  Netherlands | 6 | 2 | 8
  Canada | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) by Blinded Independent Central Review (BICR) Assessment
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of disease progression or death (whichever occurred first) according to BICR using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Disease progression was defined as an increase of greater than 20% in the sum of the longest diameter (LD) of target lesions and a 5 mm absolute increase, taking as a reference the smallest sum LD recorded since the baseline assessment or the appearance of new non-target lesions. PFS was estimated using Kaplan-Meier estimate.
Time Frame: Up to 42.8 months
Population: The ITT Population included all participants who were randomized, regardless of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 272 | 271
months | 5.5 [4.2 to 6.9] | 4.0 [3.0 to 4.4]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p = 0.0001, Log Rank — Stratified log-rank test and stratified Cox regression adjusted for stratification factors: prior chemotherapy regimens for metastatic disease, presence of visceral metastasis and endocrine therapy in the metastatic setting for at least 6 months; Hazard Ratio (HR) = 0.653, 95% CI 2-sided [0.526 to 0.812]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. OS was estimated using Kaplan-Meier estimate. Participants without documentation of death were censored on the date they were last known to be alive.
Time Frame: Up to 42.8 months
Population: Participants in the ITT Population were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 272 | 271
months | 14.5 [13.0 to 16.0] | 11.2 [10.2 to 12.6]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p = 0.0133, Log Rank — Stratified log-rank test and stratified Cox regression adjusted for stratification factors: prior chemotherapy regimens for metastatic disease, presence of visceral metastasis, and endocrine therapy in the metastatic setting for at least 6 months; Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.652 to 0.952]

3. Secondary Outcome: Objective Response Rate (ORR) by BICR and Local Investigator Review (LIR) Assessment
Description: ORR was defined as the percentage of participants who had the best overall response of either complete response (CR) or partial response (PR) that was confirmed at 4 weeks or later after initial response by BICR and LIR using RECIST 1.1. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; PR: ≥30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 42.8 months
Population: Participants in the ITT Population with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 272 | 271
percentage of participants
  ORR by BICR Assessment | 21.3 [16.6 to 26.7] | 14.0 [10.1 to 18.7]
  ORR by LIR Assessment | 16.5 [12.3 to 21.5] | 9.2 [6.1 to 13.3]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); ORR by BICR Assessment; Test type: Other; p = 0.0268, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.662, 95% CI 2-sided [1.058 to 2.609]
Statistical Analysis 2: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); ORR by LIR Assessment; Test type: Other; p = 0.0098, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.989, 95% CI 2-sided [1.174 to 3.369]

4. Secondary Outcome: Duration of Response (DOR) by BICR and LIR Assessment
Description: DOR was defined as the time from the date a response of CR or PR was first documented until the date of the first documentation of disease progression or date of death (whichever occurred first). DOR was analyzed based on both BICR and LIR assessments. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; PR: ≥30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Disease progression was defined as an increase of greater than 20% in the sum of the LD of target lesions and a 5 mm absolute increase, taking as a reference the smallest sum LD recorded since the baseline assessment or the appearance of new non-target lesions. DOR was estimated using Kaplan-Meier estimate.
Time Frame: Up to 42.8 months
Population: Participants in the ITT Population with confirmed objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 58 | 38
months
  DOR by BICR Assessment | 8.1 [6.7 to 8.9] | 5.6 [3.8 to 7.9]
  DOR by LIR Assessment: number analyzed (Participants) | 45 | 25
  DOR by LIR Assessment | 7.0 [5.6 to 8.9] | 4.3 [4.2 to 6.1]

5. Secondary Outcome: Clinical Benefit Rate (CBR) by BICR and LIR Assessment
Description: CBR was defined as the percentage of participants with the best overall response of CR, PR, or durable stable disease (duration of SD ≥ 6 months after randomization). CBR was analyzed based on both BICR and LIR assessments. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; PR: ≥30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started. PD: Disease progression was defined as an increase of greater than 20% in the sum of the LD of target lesions and a 5 mm absolute increase, taking as a reference the smallest sum LD recorded since the baseline assessment or the appearance of new non-target lesions.
Time Frame: Up to 42.8 months
Population: Participants in the ITT Population with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 272 | 271
percentage of participants
  CBR by BICR Assessment | 33.8 [28.2 to 39.8] | 22.1 [17.3 to 27.6]
  CBR by LIR Assessment | 32.4 [26.8 to 38.3] | 21.0 [16.3 to 26.4]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); CBR by BICR Assessment; Test type: Other; p = 0.0025, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.796, 95% CI 2-sided [1.227 to 2.628]
Statistical Analysis 2: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); CBR by LIR Assessment; Test type: Other; p = 0.0024, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.834, 95% CI 2-sided [1.237 to 2.717]

6. Secondary Outcome: PFS by LIR Assessment
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of disease progression or death (whichever occurred first) according to LIR using RECIST 1.1. Disease progression was defined as an increase of greater than 20% in the sum of the LD of target lesions and a 5 mm absolute increase, taking as a reference the smallest sum LD recorded since the baseline assessment or the appearance of new non-target lesions. PFS was estimated using Kaplan-Meier estimate.
Time Frame: Up to 42.8 months
Population: Participants in the ITT Population were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 272 | 271
months | 4.3 [3.8 to 5.4] | 3.1 [2.7 to 4.0]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p = 0.0010, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.728, 95% CI 2-sided [0.602 to 0.881]

7. Secondary Outcome: Time to Deterioration (TTD) of Global Health Status/Quality of Life (QoL) Scale as Measured by European Organization for Research and Treatment of Cancer Quality of Life for Cancer Patients, Core Questionnaire Version 3.0 (EORTC QLQ-C30)
Description: TTD was defined as the time from randomization to the first date a subject achieves 10-point deterioration from baseline in the global health status/QoL scale.The EORTC QLQ-C30 is a 30-item questionnaire to assess QoL of cancer patients. It has 5 functional scales(physical,role,emotional,cognitive, social)1 global health status scale,3 symptom scales (fatigue, nausea and vomiting, pain),and 6 single items(dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties). Participant responses to global health status,'How would you rate your overall health during the past week?' (Item 29)and the QoL 'How would you rate your overall quality of life during the past week?'(Item 30)questions were scored on 7-point scale (1=very poor; 7=excellent). All scales and single-item measures range in score from 0 to 100. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100. Higher scores for GHS show a better level of functioning.
Time Frame: Up to 37.8 months
Population: The HRQOL-Evaluable Population included all participants who had an evaluable assessment at baseline and at least 1 evaluable assessment at postbaseline visits. Participants with a baseline global health status/QOL score ≥ 10 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 234 | 207
months | 4.3 [3.1 to 5.7] | 3.0 [2.2 to 3.9]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p = 0.0059, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.612 to 0.922]

8. Secondary Outcome: TTD of Pain Score as Measured by EORTC QLQ-C30
Description: TTD was defined as the time from randomization to the first date a subject achieves 10-point deterioration from baseline in the pain score.The EORTC QLQ-C30 is a questionnaire to assess quality of life, it is composed of 30 questions(items) resulting in 5 functional scales(physical, role, emotional, cognitive, social),1 global health status scale,3 symptom scales (fatigue, nausea and vomiting, pain),and 6 single items(dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties). All of the scales and single-item measures range in score from 0 to 100. Participant responses to 2 questions about pain, 'Have you had pain' and 'Did pain interfere with your daily activities' were scored on 4-point scale (1=not at all;4=very much). Summed raw scores were standardized by linear transformation so that scores ranges from 0 to 100. Higher scores on the symptom scales indicate a higher level of symptoms (i.e. a worse state of the participant).
Time Frame: Up to 37.8 months
Population: Participants in the HRQOL-Evaluable Population with baseline pain score ≤ 90 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 229 | 202
months | 3.8 [2.8 to 5.0] | 3.5 [2.8 to 5.0]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p = 0.4151, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.748 to 1.126]

9. Secondary Outcome: TTD of Fatigue Score as Measured by EORTC QLQ-C30
Description: TTD was defined as the time from randomization to the first date a subject achieves 10-point deterioration from baseline in the fatigue score.The EORTC QLQ-C30 is a questionnaire to assess quality of life, it is composed of 30 questions(items) resulting in 5 functional scales(physical, role, emotional, cognitive, social),1 global health status scale,3 symptom scales (fatigue, nausea and vomiting, pain),and 6 single items(dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties).All of the scales and single-item measures range in score from 0 to 100.Participant responses to 3 questions about fatigue 'Did you need to rest', 'Have you felt weak' and 'Were you tired' were scored on a 4-point scale (1=not at all;4=very much).Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100. Higher scores on the symptom scales indicate a higher level of symptoms (i.e. a worse state of the participant).
Time Frame: Up to 37.8 months
Population: Participants in the HRQOL-Evaluable Population with baseline fatigue score ≤ 90 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 234 | 205
months | 2.2 [1.6 to 2.8] | 1.4 [1.1 to 1.9]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p = 0.0021, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.732, 95% CI 2-sided [0.598 to 0.894]

10. Secondary Outcome: Percentage of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a subject administered a medicinal product that does not necessarily have a causal relationship with this treatment. TEAEs were defined as any AEs that begin or worsen on or after the start of study drug through 30 days after the last dose of the study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0.
Time Frame: Up to 43.4 months
Population: The Safety Population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 268 | 249
percentage of participants | 100.0 | 96.0

11. Secondary Outcome: Percentage of Participants Who Experienced Treatment Emergent Serious Adverse Events (TESAEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0. An AE that met one or more of the following outcomes was classified as serious:
  * Fatal
  * Life-threatening
  * Disabling/incapacitating
  * Results in hospitalization or prolongs a hospital stay
  * A congenital abnormality
  * Other important medical events may also be considered serious AEs if they may require medical or surgical intervention to prevent one of the outcomes listed above
Time Frame: Up to 43.4 months
Population: Participants in the Safety Population were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 268 | 249
percentage of participants | 27.6 | 19.3

12. Secondary Outcome: Percentage of Participants Who Experienced the Worst Laboratory Abnormalities Grade 3 or 4 Post-Baseline
Description: Blood samples were collected for hematology, serum chemistry, and the laboratory abnormalities were assessed. A treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from baseline at any time postbaseline up to and including the date of last study drug dose plus 30 days.The most severe graded abnormality observed post-baseline for each graded test was counted for each participant. Safety as assessed by grading of laboratory values and AEs according to the National Cancer Institutes' Common Terminology Criteria for Adverse Events (NCI CTCAE) covering grades 0-5 (0=Normal, 1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening, 5=Death). The percentage of participants with worst postbaseline grades 3 or 4 are reported.
Time Frame: Up to 43.4 months
Population: Participants in the Safety Population with post-baseline values were analyzed. 'Number Analyzed' indicates participants with post-baseline values with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 265 | 242
percentage of participants
  Alanine Aminotransferase Increased: number analyzed (Participants) | 264 | 237
  Alanine Aminotransferase Increased | 1.1 | 2.1
  Hypoalbuminemia: number analyzed (Participants) | 262 | 236
  Hypoalbuminemia | 0 | 0.4
  Alkaline Phosphatase Increased: number analyzed (Participants) | 263 | 237
  Alkaline Phosphatase Increased | 0 | 0.8
  Aspartate Aminotransferase Increased: number analyzed (Participants) | 264 | 237
  Aspartate Aminotransferase Increased | 1.5 | 1.3
  Bilirubin Increased: number analyzed (Participants) | 264 | 237
  Bilirubin Increased | 2.3 | 0.8
  Creatinine Increased: number analyzed (Participants) | 263 | 237
  Creatinine Increased | 0.4 | 1.7
  Creatinine Clearance Decreased: number analyzed (Participants) | 263 | 237
  Creatinine Clearance Decreased | 2.3 | 1.3
  Hypoglycemia: number analyzed (Participants) | 262 | 237
  Hypoglycemia | 1.1 | 0.8
  Hypermagnesemia: number analyzed (Participants) | 260 | 233
  Hypermagnesemia | 0.4 | 0
  Hypomagnesemia: number analyzed (Participants) | 260 | 233
  Hypomagnesemia | 0.8 | 0
  Hyperkalemia: number analyzed (Participants) | 263 | 237
  Hyperkalemia | 1.9 | 0
  Hypokalemia: number analyzed (Participants) | 263 | 237
  Hypokalemia | 4.2 | 0.4
  Hyponatremia: number analyzed (Participants) | 263 | 237
  Hyponatremia | 0.8 | 0.4
  Anemia: number analyzed (Participants) | 265 | 241
  Anemia | 7.5 | 5.0
  Hemoglobin Increased: number analyzed (Participants) | 265 | 241
  Hemoglobin Increased | 1.1 | 0
  Leukocytes Decreased: number analyzed (Participants) | 265 | 241
  Leukocytes Decreased | 38.9 | 25.7
  Leukocytosis: number analyzed (Participants) | 265 | 241
  Leukocytosis | 0.4 | 0.4
  Lymphocytes Decreased: number analyzed (Participants) | 265 | 241
  Lymphocytes Decreased | 21.5 | 13.7
  Lymphocytes Increased: number analyzed (Participants) | 265 | 241
  Lymphocytes Increased | 1.9 | 2.1
  Neutrophils Decreased: number analyzed (Participants) | 265 | 241
  Neutrophils Decreased | 53.2 | 40.2
  Platelets Decreased: number analyzed (Participants) | 265 | 241
  Platelets Decreased | 1.9 | 3.7

13. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) - Shift From Baseline Value to Best Value During Treatment
Description: ECOG performance status (PS) measured on-therapy assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease performance without restriction;1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature;2=Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours;3=Capable of only limited self-care;confined to bed or chair more than 50% of waking hours;4=Completely disabled; cannot carry on any self-care; totally confined to bed or chair;5=Dead. Lower score indicated good performance status. Percentage of participants with Baseline ECOG PS score and corresponding changes to the best values post-baseline have been reported.
Time Frame: Up to 43.4 months
Population: Participants in the Safety Population were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 268 | 249
percentage of participants
  Baseline ECOG 0, During Treatment ECOG 0 | 34.9 | 38.7
  Baseline ECOG 0, During Treatment ECOG 1 | 7.8 | 8.9
  Baseline ECOG 0, During Treatment ECOG 2 | 0 | 0.4
  Baseline ECOG 1, During Treatment ECOG 0 | 19.4 | 11.5
  Baseline ECOG 1, During Treatment ECOG 1 | 36.4 | 38.3
  Baseline ECOG 1, During Treatment ECOG 2 | 1.6 | 2.1

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality: Up to 43.4 months
Description: Adverse Events: The Safety Population included all participants who received at least 1 dose of study drug; All-Cause Mortality: The ITT Population included all participants who were randomized, regardless of whether they received study treatment or not.
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
All-Cause Mortality (participants affected / at risk) | 234/272 | 238/271
Serious Adverse Events (participants affected / at risk) | 74/268 | 48/249
Other Adverse Events (participants affected / at risk) | 264/268 | 234/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan (N=268) | Treatment of Physician's Choice (TPC) (N=249)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 10
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0
Blepharospasm (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 5
Neutropenic colitis (Gastrointestinal disorders) | 5 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0
Covid-19 pneumonia (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 5
Pyelonephritis (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 2 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Urosepsis (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device leakage (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Embolism (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan (N=268) | Treatment of Physician's Choice (TPC) (N=249)
Anaemia (Blood and lymphatic system disorders) | 97 | 68
Leukopenia (Blood and lymphatic system disorders) | 37 | 25
Lymphopenia (Blood and lymphatic system disorders) | 32 | 29
Neutropenia (Blood and lymphatic system disorders) | 184 | 134
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 41
Abdominal distension (Gastrointestinal disorders) | 17 | 8
Abdominal pain (Gastrointestinal disorders) | 51 | 34
Abdominal pain upper (Gastrointestinal disorders) | 26 | 15
Constipation (Gastrointestinal disorders) | 93 | 61
Diarrhoea (Gastrointestinal disorders) | 163 | 57
Dry mouth (Gastrointestinal disorders) | 16 | 5
Dyspepsia (Gastrointestinal disorders) | 19 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 9
Nausea (Gastrointestinal disorders) | 157 | 86
Stomatitis (Gastrointestinal disorders) | 23 | 18
Vomiting (Gastrointestinal disorders) | 63 | 39
Asthenia (General disorders) | 62 | 49
Fatigue (General disorders) | 106 | 81
Mucosal inflammation (General disorders) | 23 | 14
Oedema peripheral (General disorders) | 17 | 14
Pain (General disorders) | 14 | 11
Pyrexia (General disorders) | 38 | 44
Urinary tract infection (Infections and infestations) | 24 | 24
Alanine aminotransferase increased (Investigations) | 30 | 37
Aspartate aminotransferase increased (Investigations) | 34 | 44
Blood alkaline phosphatase increased (Investigations) | 25 | 27
Blood bilirubin increased (Investigations) | 8 | 14
Blood lactate dehydrogenase increased (Investigations) | 9 | 13
Weight decreased (Investigations) | 15 | 14
Decreased appetite (Metabolism and nutrition disorders) | 57 | 52
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 30 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 30
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 13
Dizziness (Nervous system disorders) | 23 | 10
Headache (Nervous system disorders) | 44 | 36
Neuropathy peripheral (Nervous system disorders) | 11 | 20
Paraesthesia (Nervous system disorders) | 8 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 16
Insomnia (Psychiatric disorders) | 21 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 38
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 128 | 46
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 6
Rash (Skin and subcutaneous tissue disorders) | 24 | 14
Hypertension (Vascular disorders) | 16 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03901339/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03901339/SAP_001.pdf